CLINICAL TRIAL: NCT01513083
Title: A Phase I, Open Label, Parallel Group, Pharmacokinetic Study of Trastuzumab Emtansine in Patients With HER2-Positive Metastatic Breast Cancer and Normal or Reduced Hepatic Function
Brief Title: A Study of Trastuzumab Emtansine in Patients With HER2-Positive Metastatic Breast Cancer and Normal or Reduced Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO25499; 2011-004591-10 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (3):
- Mild hepatic dysfunction (Experimental)
  Interventions: Drug: trastuzumab emtansine
- Moderate hepatic dysfunction (Experimental)
  Interventions: Drug: trastuzumab emtansine
- Normal hepatic function (Experimental)
  Interventions: Drug: trastuzumab emtansine

INTERVENTIONS:
Drug: trastuzumab emtansine — Multiple intravenous doses

SUMMARY:
This open-label, parallel group study will evaluate the pharmacokinetics and safety of trastuzumab emtansine in patients with HER2-positive metastatic breast cancer and normal or reduced hepatic function. Patients will receive trastuzumab emtansine intravenously on Day 1 of each 3-week cycle. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically documented invasive metastatic breast cancer
* Human epidermal growth factor receptor 2 (HER2) -positive disease
* Adequate bone marrow and organ function (other than hepatic dysfunction allowed by protocol)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Left ventricular ejection fraction >/=50%
* Normal hepatic function, or mild to moderate hepatic impairment (Child-Pugh Class A or B)

Exclusion Criteria:

* History of Grade >/=3 infusion reaction, hypersensitivity reaction, or pneumonitis in response to trastuzumab
* Investigational therapy or any other anticancer therapy </=28 days before first study treatment
* Previous treatment with trastuzumab emtansine
* Brain metastases that are untreated or symptomatic or require therapy to control symptoms or any radiation, surgery or other therapy to control symptoms from brain metastases within 1 month of the first study treatment
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above
* Current peripheral neuropathy of Grade >/=2
* Child-Pugh Class C hepatic impairment
* Encephalopathy >/= Grade 2
* For patients with normal hepatic function: history of drug or alcohol addiction or history of hepatitis B and/or hepatitis C
* Active hepatitis A, B and/or C
* Current unstable ventricular arrhythmia requiring treatment
* History of symptomatic CHF (NYHA Classes II-IV)
* History of myocardial infarction or unstable angina within 6 months of enrollment
* History of a decrease in LVEF to<40% or symptomatic CHF with previous trastuzumab treatment
* Pregnant or lactating women
* Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve | Multiple sampling pre- and up to 21 days post-dose Cycles 1-3

SECONDARY OUTCOMES:
Safety: Incidence of adverse events in patients with mild or moderate hepatic impairment as compared to patients with normal hepatic function | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (4):
  - Fort Myers, Florida
  - Detroit, Michigan
  - Portland, Oregon
  - Nashville, Tennessee
- Canada (2):
  - Ottawa, Ontario
  - Toronto, Ontario
- France (3):
  - Marseille
  - Paris
  - Toulouse
- Italy (2):
  - Catanzaro, Calabria
  - Udine, Friuli Venezia Giulia
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid